CLINICAL TRIAL: NCT00407758
Title: A Phase II Evaluation of Enzastaurin (Lilly IND # 60, 933) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Enzastaurin in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170J; CDR0000517318; LILLY-H6Q-MC-S025
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Drug: enzastaurin hydrochloride

SUMMARY:
RATIONALE: Enzastaurin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well enzastaurin works in treating patients with persistent or recurrent ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy of enzastaurin hydrochloride, in terms of 6-month progression-free survival or objective tumor response, in patients with recurrent or persistent ovarian epithelial or primary peritoneal cancer.
* Determine the nature and degree of toxicity of this regimen in these patients.

Secondary

* Determine the duration of progression-free and overall survival of patients treated with this regimen.
* Determine the effects of prognostic variables, including platinum sensitivity, initial performance status, and age, in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral enzastaurin hydrochloride 3 times on day 1 and then once daily on days 2-28 of course 1. For all subsequent courses, patients receive enzastaurin hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 68 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma
* Recurrent or persistent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Must have ≥ 1 target lesion to assess response

    * Tumors within a previously irradiated field are designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence ≥ 90 days after completion of radiotherapy
* Must have received 1 prior platinum-based chemotherapy regimen containing carboplatin, cisplatin, or another organoplatinum compound for management of primary disease

  * Initial treatment may have included high-dose therapy, consolidation therapy, or extended therapy administered after surgical or nonsurgical assessment
  * Must meet any 1 of the following criteria for platinum-based therapy:

    * Disease progression during therapy
    * Treatment-free interval after completion of treatment < 12 months
    * Disease persistence after completion of therapy
* Ineligible for a higher priority GOG clinical trial

PATIENT CHARACTERISTICS:

* GOG performance status 0-1 (for patients who received 2 prior treatment regimens) OR 0-2 (for patients who received 1 prior treatment regimen)
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL (transfusions allowed)
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* Alkaline phosphatase ≤ 3 times ULN (5 times ULN if liver metastases are present)
* AST and ALT ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to swallow tablets
* No sensory or motor neuropathy > grade 1
* No active infection requiring antibiotics
* No other invasive malignancies or evidence of cancer within the past 5 years except nonmelanoma skin cancer
* No serious systemic disorders that would preclude study compliance, including an abnormal ECG indicative of cardiac disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior anticancer hormonal therapy
* No more than 1 additional cytotoxic regimen for management of recurrent or persistent disease
* At least 4 weeks since other prior anticancer therapy, including immunotherapy
* At least 30 days since prior investigational drugs
* No prior enzastaurin hydrochloride
* No prior radiotherapy to > 25% of marrow-bearing areas
* No prior noncytotoxic therapy, including bevacizumab, for recurrent or persistent disease
* No prior treatment that would preclude treatment on this protocol
* No concurrent chemotherapy, immunotherapy, or other experimental medications
* No concurrent enzyme-inducing antiepileptic drugs, including carbamazepine, phenobarbital, or phenytoin
* No other concurrent systemic anticancer therapy
* No concurrent radiotherapy, including palliative radiotherapy
* No concurrent agents that stimulate thrombopoiesis
* No concurrent amifostine or other protective reagents
* Concurrent hormone replacement therapy allowed
* Concurrent bisphosphonates allowed provided bony metastases are present

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Usha, MD, Study Chair — Rush University Medical Center; Jean A. Hurteau, MD, Study Chair — Endeavor Health
Locations (16):
- United States (16):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Usha L, Sill MW, Darcy KM, Benbrook DM, Hurteau JA, Michelin DP, Mannel RS, Hanjani P, De Geest K, Godwin AK. A Gynecologic Oncology Group phase II trial of the protein kinase C-beta inhibitor, enzastaurin and evaluation of markers with potential predictive and prognostic value in persistent or recurrent epithelial ovarian and primary peritoneal malignancies. Gynecol Oncol. 2011 Jun 1;121(3):455-61. doi: 10.1016/j.ygyno.2011.02.013. Epub 2011 Mar 17. PMID 21414654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on November 6, 2006 and was closed to accrual on May 7, 2007.
Groups:
- Enzastaurin: Loading dose of Enzastaurin 375 mg TID within 30 minutes after each meal on Day 1 followed by continuous treatment with Enzastaurin 500 mg daily within 30 minutes after the same largest meal until disease progression or adverse effects prohibit further therapy. One cycle = 28 days.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 28
Completed (Eligible and treated patients.) | 27
Not Completed | 1
Not completed — ineligible -improper prior treatment | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 4
  50-59 years | 10
  60-69 years | 6
  70-79 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above.
Time Frame: CT scan or MRI if used to follow lesions for measurable disease every other cycle for the first 6 months; every 6 months thereafter until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Partial response | 2
  Complete response | 0

2. Primary Outcome: Progression-free Survival > 6 Months Using RECIST 1.0
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for first 6 months; every 6 months thereafter until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  PFS> 6 months - Yes | 3
  PFS>6months - No | 24

3. Primary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Anemia | 1
  Constitutional | 5
  Gastrointestinal | 11
  Infection | 2
  Metabolic | 4
  Other Neurological | 1
  Pain | 5
  Pulmonary | 5
  Vascular | 1
  Death, not CTC coded | 3

4. Secondary Outcome: Duration Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
months | 15.1 [6.5 to NA] — Upper limit not yet reached

5. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
months | 1.8 [1.5 to 2.7]

6. Secondary Outcome: Prognostic Factor - Number of Patients With Platinum Sensitivity
Description: Platinum sensitive = a platinum-free interval between 6 and 12 months.
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Platinum Sensitive | 11
  Not Platinum Sensitive | 16

7. Secondary Outcome: Prognostic Factor - Initial Performance Status
Description: Performance status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Performance Status = 0 | 16
  Performance Status = 1 | 11

8. Secondary Outcome: Prognostic Factor - Age at Study Entry
Time Frame: Baseline
Population: Eligible and treated patients
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
years | 59 [53 to 71]

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 12/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzastaurin (N=27)
Death No Ctcae Term - Disease Progression Nos (General disorders) | 3
Obstruction, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzastaurin (N=27)
Rhinitis (Immune system disorders) | 4
Neutrophils (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 3
Leukocytes (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 19
Palpitations (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Sweating (General disorders) | 2
Weight Gain (General disorders) | 1
Fever (General disorders) | 1
Weight Loss (General disorders) | 1
Fatigue (General disorders) | 20
Insomnia (General disorders) | 4
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Decubitus (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Diabetes (Endocrine disorders) | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 4
Ileus (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 3
Taste Alteration (Gastrointestinal disorders) | 2
Incontinence, Anal (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 3
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Anorexia (Gastrointestinal disorders) | 12
Dehydration (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 13
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Petechiae (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Pleura (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Colon (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 5
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Vulva (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 8
Edema: Head And Neck (Blood and lymphatic system disorders) | 1
Ast (Metabolism and nutrition disorders) | 2
Gfr (Metabolism and nutrition disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alt (Metabolism and nutrition disorders) | 1
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Mood Alteration - Depression (Nervous system disorders) | 2
Mood Alteration - Anxiety (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Neuropathy-Sensory (Nervous system disorders) | 1
Neuropathy-Motor (Nervous system disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Breast (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Head/Headache (General disorders) | 3
Pain: Extremity-Limb (General disorders) | 1
Pain: Joint (General disorders) | 3
Pain: Bone (General disorders) | 1
Pain: Rectum (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 11
Pain: Tumor (General disorders) | 1
Pain: Muscle (General disorders) | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Urinary Color Change (Renal and urinary disorders) | 3
Vaginal Dryness (Reproductive system and breast disorders) | 1
Flu-Like Syndrome (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less